CLINICAL TRIAL: NCT03830554
Title: Effect of Atlas Cedarwood Essential Oil Aromatherapy on Sleep Quality Among Patients With Coronary Heart Disease: a Randomized Controlled Trial
Brief Title: Effect of Atlas Cedarwood Essential Oil Aromatherapy on Sleep Quality Among Patients With Coronary Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rawan Alghzawi (Other)
Collaborators: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor-Investigator, Rawan Alghzawi, master student at nursing faculty, Jordan University of Science and Technology
Organization: Jordan University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 15/Clinical/18
Record Dates: First submitted 2019-01-10; First posted 2019-02-05 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Sleep Quality; Coronary Heart Disease
Keywords: sleep disturbances; Aromatherapy; sleep quality; Atlas cedar wood essential oil
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Coronary Disease; Parasomnias | interventions — Aromatherapy

STUDY DESIGN:
Intervention Model Description: 96 CHD participants were approached to participate in this RCT. out of those, 22 participants reported good sleep quality (PSQI SCORE <5), their participation finished at phase one. The rest 74 participants reported poor sleep quality (PSQI score =>5) were randomly assigned either to intervention or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): product name: organic Atlas cedar wood essential oil (Cedrus Atlantica): the intervention group smell 2 drops of organic Atlas cedar wood essential oil (applied on cotton ball) for a period of five consecutive nights (at least 8 hours each night).
  Interventions: Other: Organic Atlas cedar wood essential oil (Cedrus Atantica)
- control group (No Intervention): participants of this group received no intervention.

INTERVENTIONS:
Other: Organic Atlas cedar wood essential oil (Cedrus Atantica) — At first day of admission, Intervention group received an intervention kit consist of 5 small glass essential oil bottles. Each essential oil bottle contains a small cotton ball saturated with two drops of Organic Atlas cedar wood essential oil (Cedrus Atantica). Participants were asked to open the bottle, inhale the smell directly and put it opened at 20 cm beside bed during night.
  Other Names: aromatherapy
  Arms: intervention group

SUMMARY:
Sleep-wake disturbances were found to be a common problem among patients with CHD either earlier during hospitalization or/ and after discharge Although there is an evidence that sleep-wake disturbanes occur in high rate among patients with CHD little was found about assessment and management of this problem. This randomized controlled study will assess sleep quality of stable CHD patients who were admitted for undergoing coronary angiography electively. Then it will test the hypothesis that atlas cedar wood essential oil aromatherapy have a positive effect on sleep quality of CHD patients.

DETAILED DESCRIPTION:
The primary aim is testing the effect of Atlas cedar wood essential oil aromatherapy on sleep quality of patients after CHD.

The secondary aim is estimating the prevalence of sleep-wake disturbances (difficulty falling asleep, staying asleep, inadequate sleep duration, dissatisfaction with a sleep and excessive daytime sleepiness) among recruited CHD patients.

- data were collected by two phase:

* phase one: sleep quality of recruited CHD patients, who were admitted for undergoing coronary angiography electively, were assessed using Pittsburg Sleep Quality Index (PSQI). CHD participants who were reported poor sleep quality (=>5) in PSQI score will randomly allocated by toss either to intervention or control group.
* Phase two:

  1. Intervention group received an atlas cedar wood aromatherapy for five consecutive nights.
  2. Control group received no intervention.
  3. Sleep quality of both group participants re-assessed at second day and six day of recruitment, respectively, using PSQI.

ELIGIBILITY:
Inclusion Criteria:

1. stable CHD patients with history of myocardial infarction, stable angina, unstable angina or acute coronary syndrome who were admitted for elective coronary angiograph (cardiac catheterization) during the study period.
2. age of participants must be between 20-64 years old.
3. participants must have an ability to understand and communicate with the researchers.

Exclusion Criteria:

included CHD patient were excluded if they:

1. pregnant women or who has a plan for pregnancy as well as any patients who their care giver is pregnant
2. have a recent cardiac attack within 24-48 hours or had a history or risk of heart failure or cardiogenic shock were excluded.
3. have problems in smell sensations , history of breathing difficulties and disorders such as asthma, sleep apnea or allergies to plants and flowers parts were excluded, too.
4. have history of psychological disorders (i.e., depression) or psychiatric disorders (i.e., schizophrenia) were excluded
5. using prescribed sedatives drugs or other complementary therapy likes herbal remediates or even aromatherapy in recent one week were excluded
6. shift workers.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2018-11-05 (Actual)

PRIMARY OUTCOMES:
Demographic and Situational Data Sheet | at the day of admission
  The participants were asked to fill a demographic and situational data sheet that is bulit by the researches based on the inclusion and exclusion criteria of the study. this sheet assess participants' age, gender, marital status, educational level, occupation and bed time habits. Also it have a disease related questions, that consists of time of diagnosis of CHD, presence of other chronic disease (physiological or psychological disease), previous complaint of sleep problem, medication history rather than used for CHD treatments, using of complementary therapy with justification.Through this data, female participants were asked if they are in menopausal period, pregnant or have a plan of pregnancy during next month.
sleep quality score during past month before admission using Arabic version of PITTSBURGH SLEEP QUALITY INDEX (PSQI) | during past month before admission
  sleep quality (during past month) of participants was assessed at the day of each patient admission. Arabic version of PITTSBURGH SLEEP QUALITY INDEX is a valid and reliable version of original English version that is a self-rated questionnaire used for measuring sleep quality for duration of one month interval. The instrument consists of 24 questions (19 self-rated questions and 5 questions measures objective sleep quality from bed partner. Self- rated question are combined to form seven component score. Each component has a score range from 0 point (no difficulty) to 3 point (extreme difficulty). Global PSQI score results from summation of seven component scores. It have a range from 0 point (no difficulty in all area) to 21 points (severe difficulties in all area). Global PSQI score >=5 indicate a poor sleep quality where a total score <5 indicate a good sleep quality.
sleep quality score during past day of hospitalization (before undergoing cardiac catheterization) using Arabic version of PITTSBURGH SLEEP QUALITY INDEX (PSQI) | one day during hospitalization
  sleep quality of participants was assessed for the second time after sleeping one night in hospital using Arabic version of PITTSBURGH SLEEP QUALITY INDEX (one day used instead of month words). Arabic version of PITTSBURGH SLEEP QUALITY INDEX is a valid and reliable version of original English version that is a self-rated questionnaire. The instrument consists of 24 questions (19 self-rated questions and the rest 5 questions are measured objective sleep quality from bed partner. Self- rated question are only used in the scoring and they are combined to form seven component score. Each component has a score range from 0 point (no difficulty) to 3 point (extreme difficulty). Global PSQI score results from summation of seven component scores. It have a range from 0 point (no difficulty in all area) to 21 points (severe difficulties in all area). Global PSQI score >=5 indicate a poor sleep quality where total score <5 indicate a good sleep quality.
sleep quality score during past five days (after undergoing cardiac catheterization) using Arabic version of PITTSBURGH SLEEP QUALITY INDEX | five days after admission
  sleep quality of participants was assessed for the third time after five days from admission using Arabic version of PITTSBURGH SLEEP QUALITY INDEX (five days was used instead of month words in original tool). Arabic version of PITTSBURGH SLEEP QUALITY INDEX is a valid and reliable version of original English version that is a self-rated questionnaire. The instrument consists of 24 questions (19 self-rated questions and the rest 5 questions are measured objective sleep quality from bed partner. Self- rated question are only used in the scoring and they are combined to form seven component score. Each component has a score range from 0 point (no difficulty) to 3 point (extreme difficulty). Global PSQI score results from summation of seven component scores. It have a range from 0 point (no difficulty in all area) to 21 points (severe difficulties in all area). Global PSQI score >=5 indicate a poor sleep quality where total score <5 indicate a good sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: rawan algzawy, Principal Investigator — Dean of graduate studies at Jordan university of science and Technology; wejdan khater, Study Director — Dean of graduate studies at Jordan university of science and Technology
Locations (1):
- ordan University of Science and Technology, Irbid, Al-ramtha, Jordan

REFERENCES:
- [Background] Sano A, Sei H, Seno H, Morita Y, Moritoki H. Influence of cedar essence on spontaneous activity and sleep of rats and human daytime nap. Psychiatry Clin Neurosci. 1998 Apr;52(2):133-5. doi: 10.1111/j.1440-1819.1998.tb00991.x. PMID 9628112
- [Background] Michal M, Wiltink J, Kirschner Y, Schneider A, Wild PS, Munzel T, Blettner M, Schulz A, Lackner K, Pfeiffer N, Blankenberg S, Tschan R, Tuin I, Beutel ME. Complaints of sleep disturbances are associated with cardiovascular disease: results from the Gutenberg Health Study. PLoS One. 2014 Aug 5;9(8):e104324. doi: 10.1371/journal.pone.0104324. eCollection 2014. PMID 25093413
- [Background] Martins DF, Emer AA, Batisti AP, Donatello N, Carlesso MG, Mazzardo-Martins L, Venzke D, Micke GA, Pizzolatti MG, Piovezan AP, dos Santos AR. Inhalation of Cedrus atlantica essential oil alleviates pain behavior through activation of descending pain modulation pathways in a mouse model of postoperative pain. J Ethnopharmacol. 2015 Dec 4;175:30-8. doi: 10.1016/j.jep.2015.08.048. Epub 2015 Sep 4. PMID 26344850
- [Background] Khaled, S., Lourance, A.-H., & Ahmad, D. (2012). Psychometric testing of the Arabic version of the Pittsburgh Sleep Quality Index (A-PSQI) among coronary artery disease patients in Jordan. J Nat Sci Res, 2, 15-19.
- [Background] Hwang E, Shin S. The effects of aromatherapy on sleep improvement: a systematic literature review and meta-analysis. J Altern Complement Med. 2015 Feb;21(2):61-8. doi: 10.1089/acm.2014.0113. Epub 2015 Jan 13. PMID 25584799
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Alcantara C, Peacock J, Davidson KW, Hiti D, Edmondson D. The association of short sleep after acute coronary syndrome with recurrent cardiac events and mortality. Int J Cardiol. 2014 Feb 1;171(2):e11-2. doi: 10.1016/j.ijcard.2013.11.135. Epub 2013 Dec 7. No abstract available. PMID 24365609
- [Background] Ali, B., Al-Wabel, N. A., Shams, S., Ahamad, A., Khan, S. A., & Anwar, F. (2015). Essential oils used in aromatherapy: A systemic review. Asian Pacific Journal of Tropical Biomedicine, 5(8), 601-611.
- [Background] Andrechuk CR, Ceolim MF. Sleep quality and adverse outcomes for patients with acute myocardial infarction. J Clin Nurs. 2016 Jan;25(1-2):223-30. doi: 10.1111/jocn.13051. PMID 26769209
- [Background] King, L., Wright, B., & Reynolds, A. (2015). AROMATHERAPY.